CLINICAL TRIAL: NCT04886791
Title: Vaginal Hysterectomy Versus Vaginal Assisted NOTES Hysterectomy (VANH): a Randomised Controlled Trial
Brief Title: Vaginal NOTES Hysterectomy Versus Vaginal Hysterectomy
Acronym: VANH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ilse Bekkers, Doctor in training to be a gynaecologist, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL76240.096.21
Record Dates: First submitted 2021-04-26; First posted 2021-05-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hysterectomy; Natural Orifice Transluminal Endoscopic Surgery; Vaginal Hysterectomy
Keywords: NOTES surgery; vNOTES; VANH; Vaginal hysterectomy; Hysterectomy
MeSH Terms: interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Intervention Model Description: Single-blinded, multicentre, randomised controlled trial
Who Masked: Participant
Masking Description: Participant is blinded for which surgery they will undergo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VANH hysterectomy (Experimental): Access to the peritoneal cavity will be performed similar to vaginal surgery by a circular incision around the cervix, anterior and posterior colpotomy and transsecting the sacro-uterine ligaments. The vNOTES port will be placed to get access to the abdominal cavity and a pneumoperitoneum will be created. After positioning in 20o degree Trendelenburg laparoscopic instruments will be introduced. The peritoneal cavity and ureters are inspected. The hysterectomy is performed by dissecting from caudally to cranially. The fallopian tubes will be removed elective after counselling in the outpatient clinic and the ovaries will be removed on indication only. Haemostasis is checked and the vNOTES port and the uterus are removed trans-vaginally and the pneumoperitoneum is deflated. The vaginal cuff will be closed using a running Vicryl-1 suture. The urinary bladder catheter will be removed directly postoperative.
  Interventions: Procedure: Vaginal NOTES hysterectomy
- Vaginal hysterectomy (Active Comparator): A circumferential incision is made around the cervix. Access to the peritoneal cavity will be performed through anterior and posterior colpotomy. The sacro-uterine ligaments, ligamenta cardinalia uterine arteries will be clamped and dissected. Finally, the ovarian ligament, round ligament and fallopian tubes will be dissected and tied. The uterus will be removed and the vagina will be closed. The urinary bladder catheter will be removed directly postoperative.
  Interventions: Procedure: Vaginal hysterectomy

INTERVENTIONS:
Procedure: Vaginal NOTES hysterectomy — Vaginal assited NOTES hysterectomy
  Arms: VANH hysterectomy
Procedure: Vaginal hysterectomy — Vaginal hysterectomy
  Arms: Vaginal hysterectomy

SUMMARY:
Rationale: Natural orifice transluminal endoscopic surgery (NOTES) is a minimal invasive technique using the natural body orifices like stomach, oesophagus, bladder, rectum and vagina to access the human body for surgery. In 2012, the first vaginal NOTES (vNOTES) hysterectomy was performed. Potential benefits of vNOTES hysterectomy, also called the vaginal assisted NOTES hysterectomy (VANH) are no visible scars, less pain and a shorter hospital stay compared with laparoscopic hysterectomy as shown in the HALON trial. Up to now, no studies have compared the vNOTES hysterectomy with vaginal hysterectomy.

Objective: The aim of this study is to compare the vNOTES hysterectomy with the vaginal hysterectomy for same day-discharge (SDD), complications, treatment related outcomes, post-operative recovery, quality of life and cost-effectiveness.

Study design: The study concerns a single-blinded, multicentre, randomised controlled trial.

Study population: Eligible women who fulfill the inclusion criteria and will undergo a hysterectomy for benign indication.

Intervention: The study population will be randomly allocated to the VANH-group, who undergo a vaginal assisted NOTES hysterectomy (intervention group) or the vaginal hysterectomy group (control-group) and the participants will be single blinded. The pre- and postoperative care will be the same for both groups.

Main study parameters/endpoints: Primary outcome is the percentage of patients that underwent the hysterectomy as in SDD setting. A total of 41 patients should be included in the control group and a total of 83 patients in the intervention group, using an enrollment ratio of 1:2, with an alpha of 0.05 and a power of 0.8.

The secondary outcomes are complications, treatment related outcomes, post-operative recovery, quality of life and cost-effectiveness.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

vNOTES is a new surgical technique, but a combination of two existing techniques namely the vaginal hysterectomy and the laparoscopic hysterectomy. Only one randomized controlled trial has been published, comparing the total laparoscopic hysterectomy (TLH) with the VANH, which shows no inferiority of the vNOTES technique compared to a laparoscopy. A recent case series study has been published about the complication rate in VANH. There was a total complication rate in the hysterectomy group of 5.2%, in which 1.4% was intra-operative and 3.8% postoperative. Theoretically it is possible that the VANH causes less intra-operative complications because of an improved view during the procedure. No further literature is known about VH versus VANH. Participants of the study should fill in multiple questionnaires before randomization and postoperative about their general health, pain experience and used analgesics.

DETAILED DESCRIPTION:
The hysterectomy is one of the most performed gynaecological surgeries worldwide.

In the Netherlands about 14.500 hysterectomies are performed yearly. The most common benign indications to perform a hysterectomy are abnormal uterine bleeding, uterine leiomyomas, endometriosis or adenomyosis, chronic pelvic pain, uterine prolapse, benign ovarian neoplasm, hyperplasia or atypia of the endometrium or cervical dysplasia.

The four approaches to perform a hysterectomy for benign disease are abdominal hysterectomy (AH), vaginal hysterectomy (VH), (total) laparoscopic hysterectomy ((T)LH) and robotic-assisted hysterectomy (RH).

VH appears to be superior to the AH, resulting in a quicker recovery. The LH results in a quicker recovery than the AH and VH, but increases the risks of damage to the bladder or ureter. That is why a recent Cochrane review advises to perform a VH when feasible for women undergoing a hysterectomy for a benign indication. When VH is technically not feasible, a LH or AH is performed. LH resulted in more rapid recovery, fewer febrile episodes and less wound complications compared to AH. The RH is not superior compared to the LH and is associated with higher costs.

Since the introduction of laparoscopy, the VH and AH decreased and the rate of LH significantly increased between 2002 and 2012. Performing a LH gives the opportunity to inspect the abdominal cavity and to easily perform an opportunistic salpingectomy compared to VH. An opportunistic salpingectomy during a hysterectomy for benign indication might reduce the overall risk of ovarian cancer.

Additionally, patients experience less postoperative pain after a LH compared to a VH and therefore need less post-operative pain medication. Advantages of the VH compared to the LH are a shorter operation duration, no visible scars and a lower chance of dehiscence of the vaginal cuff.

In 2004, a novel approach of endoscopic surgery was described, 'Natural Orifice Transluminal Endoscopic Surgery (NOTES) by researchers at the John Hopkins University. It is a surgical technique using natural orifices of the body (e.g. mouth, anus, urethra, vagina) to perform scarless surgery. The vaginal approach is called the vNOTES technique. NOTES is an emerging field within minimal access surgery, evolves and presents multiple possibilities for innovation and development. The initial approach was trans gastric, but subsequently, NOTES has been evolved, resulting in trans rectal, trans gastric, transvaginal, and transurethral approaches nowadays.

In 2012, the first vNOTES hysterectomy, also called vaginal assisted NOTES hysterectomy (VANH) was performed. vNOTES surgery can be used for different indications, for example hysterectomy, adnexectomy or salpingectomy in case of an ectopic pregnancy.

In 2018, the first randomised controlled trial (RCT) comparing TLH with VANH in 70 women was published. This HALON trial showed VANH was non-inferior to TLH. Compared to TLH, surgery time was significantly shorter, patients experience less post-operative pain and same day discharge (SDD) was possible in 77% of the women who underwent the VANH compared to 43% after TLH. Besides, the VANH showed less post-operative complications.

Except for the HALON trial and two retrospective studies and case-control studies, there is little literature about VANH.

No studies have been performed comparing the VH with the VANH. Because the VH is the preferred method to perform a hysterectomy for a benign indication, there is a need to compare VH with VANH and to explore the indications to perform a VANH.

The aim of this study is to compare the VANH with the VH for same day discharge (SDD), complications, treatment related outcomes, post-operative recovery, quality of life and cost-effectiveness.

We hypothesize that patients who underwent a VANH procedure are more often able to be treated in SDD setting.

ELIGIBILITY:
Inclusion Criteria:

* Written and orally given informed consent
* 18 years and older
* Native Dutch speaker or in control of the Dutch language in speaking and writing
* Indication for hysterectomy for benign indication
* Possible to perform a VH judged by experienced (resident) gynaecologist during gynaecological examination

Exclusion Criteria:

* Any contra-indication for VH (for example, large uterus myomatosus, not enough descensus, etc) as judged by experienced gynaecologist
* History of more than 1 caesarean section
* History of endometriosis
* History of rectal surgery
* History of pelvic radiation
* Suspected rectovaginal endometriosis
* History of pelvic inflammatory disease, especially prior tubo-ovarian or pouch of Douglas abscess or suspected adhesions due to (ruptured) inflammatory disease (for example ruptured appendicitis)
* Virginity
* Pregnancy
* Indication for anterior or posterior colporrhaphy during the same surgery
* Indication of mid urethral slings
* Uterus myomatosus will not be an exclusion criteria but the surgeon will indicate if it is possible to remove the uterus vaginally.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 124 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of same day discharge | First 24hours after surgery
  Same day discharge

SECONDARY OUTCOMES:
Complications | Week 6 after surgery
  Severity scored by Clavien Dindo classifications
Treatment related outcomes-1 | During surgery
  Conversion
Intended number of salphingectomies in each group | During surgery
  Intended number of salphingectomies
Performed number of salphingectomies in each group | During surgery
  Performed number of salphingectomies
Recovery Index-10 (RI-10) pre- and postoperative | Week 12 after surgery
  Recovery Index-10 (RI-10)
Health- related Quality of LIfe (EQ-5D-5L questionnaire) | Week 12 after surgery
  EQ-5D-5L questionnaire
Costs | Week 12 after sugery
  Intervention costs, hospital costs, health care costs outside the hospital (using iMCQ questionnaire)
Cost effectiveness | Week 12 after surgery
  Cost effectiveness between vaginal NOTES hysterectomy versus vaginal hysterectomy comparing the costs as mentioned at outcome 8
Treatment related outcomes-2 | During surgery
  Time in operating theatre in minutes
Treatment related outcomes- 3 | During surgery
  Surgery time in minutes
Treatment related outcomes -4 | During surgery
  blood loss in mL
Treatment related outcomes -5 | First 24 hours after surgery
  Pain after surgery measured on numeric rating scale
Treatment related outcomes -6 | Day 7 after surgery
  Recovery of pain in first 7 days after surgery measured on numeric rating scale
Treatment related outcomes - 7 | Day 7 after surgery
  Use of analgesics
Treatment related outcomes - 8 | Week 6 after surgery
  resumption of daily activity
Treatment related outcomes - 9 | Week 6 after surgery
  hospital re-admission

CONTACTS AND LOCATIONS:
Overall Officials: Martine Wassen, Principal Investigator — Zuyderland Medical Centre
Locations (2):
- Netherlands (2):
  - Catharina Medical Centre, Eindhoven, North Brabant
  - Zuyderland Medical Centre, Heerlen, North Brabant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baekelandt J, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BW, Bosteels JJ. Authors' reply re: Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery versus laparoscopy as a daycare procedure: a randomised controlled trial. BJOG. 2019 Jul;126(8):1078-1079. doi: 10.1111/1471-0528.15744. Epub 2019 Apr 24. No abstract available. PMID 31020729
- [Background] Baekelandt J, Kapurubandara S. Benign Gynaecological procedures by vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES): Complication data from a series of 1000 patients. Eur J Obstet Gynecol Reprod Biol. 2021 Jan;256:221-224. doi: 10.1016/j.ejogrb.2020.10.059. Epub 2020 Oct 28. PMID 33248377
- [Background] Hammer A, Rositch AF, Kahlert J, Gravitt PE, Blaakaer J, Sogaard M. Global epidemiology of hysterectomy: possible impact on gynecological cancer rates. Am J Obstet Gynecol. 2015 Jul;213(1):23-29. doi: 10.1016/j.ajog.2015.02.019. Epub 2015 Feb 25. PMID 25724402
- [Background] Committee Opinion No. 701 Summary: Choosing The Route Of Hysterectomy For Benign Disease. Obstet Gynecol. 2017 Jun;129(6):1149-1150. doi: 10.1097/AOG.0000000000002108. PMID 28538491
- [Background] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Background] Neis KJ, Zubke W, Romer T, Schwerdtfeger K, Schollmeyer T, Rimbach S, Holthaus B, Solomayer E, Bojahr B, Neis F, Reisenauer C, Gabriel B, Dieterich H, Runnenbaum IB, Kleine W, Strauss A, Menton M, Mylonas I, David M, Horn LC, Schmidt D, Gass P, Teichmann AT, Brandner P, Stummvoll W, Kuhn A, Muller M, Fehr M, Tamussino K. Indications and Route of Hysterectomy for Benign Diseases. Guideline of the DGGG, OEGGG and SGGG (S3 Level, AWMF Registry No. 015/070, April 2015). Geburtshilfe Frauenheilkd. 2016 Apr;76(4):350-364. doi: 10.1055/s-0042-104288. PMID 27667852
- [Background] Johnson N, Barlow D, Lethaby A, Tavender E, Curr L, Garry R. Methods of hysterectomy: systematic review and meta-analysis of randomised controlled trials. BMJ. 2005 Jun 25;330(7506):1478. doi: 10.1136/bmj.330.7506.1478. PMID 15976422
- [Background] Driessen SR, Baden NL, van Zwet EW, Twijnstra AR, Jansen FW. Trends in the implementation of advanced minimally invasive gynecologic surgical procedures in the Netherlands. J Minim Invasive Gynecol. 2015 May-Jun;22(4):642-7. doi: 10.1016/j.jmig.2015.01.026. Epub 2015 Feb 3. PMID 25655043
- [Background] van Lieshout LAM, Steenbeek MP, De Hullu JA, Vos MC, Houterman S, Wilkinson J, Piek JM. Hysterectomy with opportunistic salpingectomy versus hysterectomy alone. Cochrane Database Syst Rev. 2019 Aug 28;8(8):CD012858. doi: 10.1002/14651858.CD012858.pub2. PMID 31456223
- [Background] Kalloo AN, Singh VK, Jagannath SB, Niiyama H, Hill SL, Vaughn CA, Magee CA, Kantsevoy SV. Flexible transgastric peritoneoscopy: a novel approach to diagnostic and therapeutic interventions in the peritoneal cavity. Gastrointest Endosc. 2004 Jul;60(1):114-7. doi: 10.1016/s0016-5107(04)01309-4. PMID 15229442
- [Background] Santos BF, Hungness ES. Natural orifice translumenal endoscopic surgery: progress in humans since white paper. World J Gastroenterol. 2011 Apr 7;17(13):1655-65. doi: 10.3748/wjg.v17.i13.1655. PMID 21483624
- [Background] Rolanda C, Lima E, Pego JM, Henriques-Coelho T, Silva D, Moreira I, Macedo G, Carvalho JL, Correia-Pinto J. Third-generation cholecystectomy by natural orifices: transgastric and transvesical combined approach (with video). Gastrointest Endosc. 2007 Jan;65(1):111-7. doi: 10.1016/j.gie.2006.07.050. PMID 17185089
- [Background] Nieuwenhuis D, Velthuis S, Bonjer J, Sietses C. [Transanal total mesorectal excision: a new treatment option for rectal cancer]. Ned Tijdschr Geneeskd. 2014;158(6):A7054. Dutch. PMID 24495374
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; TaTME Registry Collaborative. Transanal Total Mesorectal Excision: International Registry Results of the First 720 Cases. Ann Surg. 2017 Jul;266(1):111-117. doi: 10.1097/SLA.0000000000001948. PMID 27735827
- [Background] Su H, Yen CF, Wu KY, Han CM, Lee CL. Hysterectomy via transvaginal natural orifice transluminal endoscopic surgery (NOTES): feasibility of an innovative approach. Taiwan J Obstet Gynecol. 2012 Jun;51(2):217-21. doi: 10.1016/j.tjog.2012.04.009. PMID 22795097
- [Background] Wang CJ, Huang HY, Huang CY, Su H. Hysterectomy via transvaginal natural orifice transluminal endoscopic surgery for nonprolapsed uteri. Surg Endosc. 2015 Jan;29(1):100-7. doi: 10.1007/s00464-014-3639-y. Epub 2014 Oct 1. PMID 25270610
- [Background] Yang YS, Kim SY, Hur MH, Oh KY. Natural orifice transluminal endoscopic surgery-assisted versus single-port laparoscopic-assisted vaginal hysterectomy: a case-matched study. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):624-31. doi: 10.1016/j.jmig.2014.01.005. Epub 2014 Jan 21. PMID 24462594
- [Background] Lee CL, Wu KY, Su H, Wu PJ, Han CM, Yen CF. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery (NOTES): a series of 137 patients. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):818-24. doi: 10.1016/j.jmig.2014.03.011. Epub 2014 Mar 25. PMID 24681063
- [Background] Hanstede MM, Burger MJ, Timmermans A, Burger MP. Regional and temporal variation in hysterectomy rates and surgical routes for benign diseases in the Netherlands. Acta Obstet Gynecol Scand. 2012 Feb;91(2):220-5. doi: 10.1111/j.1600-0412.2011.01309.x. PMID 22043840
- [Background] David-Montefiore E, Rouzier R, Chapron C, Darai E; Collegiale d'Obstetrique et Gynecologie de Paris-Ile de France. Surgical routes and complications of hysterectomy for benign disorders: a prospective observational study in French university hospitals. Hum Reprod. 2007 Jan;22(1):260-5. doi: 10.1093/humrep/del336. Epub 2006 Sep 1. PMID 16950826
- [Background] Kruger PF, Mehta C, Lee P. Predictors of Length of Stay After Vaginal Hysterectomy. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S246. doi: 10.1016/j.jmig.2015.08.860. Epub 2015 Oct 15. No abstract available. PMID 27679173
- [Background] Allam IS, Makled AK, Gomaa IA, El Bishry GM, Bayoumy HA, Ali DF. Total laparoscopic hysterectomy, vaginal hysterectomy and total abdominal hysterectomy using electrosurgical bipolar vessel sealing technique: a randomized controlled trial. Arch Gynecol Obstet. 2015 Jun;291(6):1341-5. doi: 10.1007/s00404-014-3571-3. Epub 2014 Dec 19. PMID 25524534
- [Background] Morton M, Cheung VYT, Rosenthal DM. Total laparoscopic versus vaginal hysterectomy: a retrospective comparison. J Obstet Gynaecol Can. 2008 Nov;30(11):1039-1044. doi: 10.1016/S1701-2163(16)32999-1. PMID 19126286
- [Background] Sesti F, Cosi V, Calonzi F, Ruggeri V, Pietropolli A, Di Francesco L, Piccione E. Randomized comparison of total laparoscopic, laparoscopically assisted vaginal and vaginal hysterectomies for myomatous uteri. Arch Gynecol Obstet. 2014 Sep;290(3):485-91. doi: 10.1007/s00404-014-3228-2. Epub 2014 Apr 8. PMID 24710800
- [Background] Liu L, Yi J, Cornella J, Butterfield R, Buras M, Wasson M. Same-Day Discharge after Vaginal Hysterectomy with Pelvic Floor Reconstruction: Pilot Study. J Minim Invasive Gynecol. 2020 Feb;27(2):498-503.e1. doi: 10.1016/j.jmig.2019.04.010. Epub 2019 Apr 10. PMID 30980994
- [Background] Wang CJ, Go J, Huang HY, Wu KY, Huang YT, Liu YC, Weng CH. Learning curve analysis of transvaginal natural orifice transluminal endoscopic hysterectomy. BMC Surg. 2019 Jul 10;19(1):88. doi: 10.1186/s12893-019-0554-0. PMID 31291917
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04886791/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04886791/ICF_001.pdf